CLINICAL TRIAL: NCT03304496
Title: Subcutaneous Administration of Nitroglycerin to Facilitate Trans-radial Access in Coronary Procedures: a Randomized Clinical Trial (NITRAD-Sub Study).
Brief Title: Subcutaneous Nitroglycerin to Facilitate Trans-radial Access.
Acronym: NITRAD-Sub
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Daniel Coutiño-Castelán, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PT-17-044
Record Dates: First submitted 2017-09-24; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: Nitroglycerin; Vasodilator Agents; Subcutaneous Injection; Radial Artery; Coronary Angiography; Cardiac Catheterization; Coronary Angioplasty; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin (Experimental): The intervention group will receive a subcutaneous "cocktail" with 0,5 ml of 500 mcg of nitroglycerin + 1 ml of 2% simple lidocaine.
  Interventions: Drug: Nitroglycerin 100 MCG/ML Injectable Solution
- Control (Placebo Comparator): The placebo group will receive a subcutaneous injection with 0,5 ml of 0,9% saline solution + 1 ml of 2% simple lidocaine.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Nitroglycerin 100 MCG/ML Injectable Solution — Previously described.
  Arms: Nitroglycerin
Drug: Saline Solution — Previously described.
  Arms: Control

SUMMARY:
Femoral artery approach to perform coronary procedures is considered the standard technique for vascular access due to optimal catheter control, lower thromboembolic complications and immediate access due to the large diameter of the artery. Trans-radial approach has been shown to reduce major bleeding complications, vascular complications related to the site of puncture, including death from all causes, and to prevent post-procedure limb rest, greater comfort for patients, immediate ambulation, early discharge and reduction of costs. Previous studies have shown that intravenous, topical and intraarterial use of nitroglycerin produces vasodilation of the radial artery. Extravascular (subcutaneous) administration of nitroglycerin is extremely effective in restoring the radial pulse, and allows adequate cannulation.

DETAILED DESCRIPTION:
Unlike femoral access, the trans-radial approach to coronary angiography requires a greater learning curve for the inexperienced interventionist, and demands a greater technical challenge than the femoral approach, which leads to a high incidence of failures and complications, mainly in the initial stages of their formation. Some explanations for procedural failure include inability for radial artery puncture, vessel tortuosity, and radial spasm. Radial spasm has been reported from 5 to 30% in experienced centers, with a decrease to 2.5% when associated with the administration of nitrate added to local anesthesia. Although radial spasm is infrequent and usually occurs once the artery is cannulated or during manipulation of the catheters, it can sometimes occur before cannulation due to multiple unsuccessful attempts to cannulate the artery, which can also produce pain in the patient.

The investigators will conduct an experimental, placebo-controlled, longitudinal, prospective, double-blind, parallel arm clinical trial. Patients will be randomized to receive 1:1 an intervention or placebo. Intervention group will receive a subcutaneous "cocktail" with 0.5 ml of 500 mcg of nitroglycerin + 1 ml of 2% simple lidocaine. Placebo group will receive a subcutaneous injection with 0.5 ml of 0.9% saline solution + 1 ml of 2% simple lidocaine.

The investigators hypothesize that the maneuver (subcutaneous infiltration of local anesthetic together with nitroglycerin) will facilitate radial access in terms of fewer punctures until the insertion of the arterial introducer, shorter access time, lower incidence of radial spasm, and lower crossover rate to femoral access, compared with placebo. In terms of safety, the investigators do not believe that the maneuver represents a risk to the patient in terms of incidence of hypotension or headache. In fact, the investigators believe that the maneuver will provide less pain at the site of puncture referred by the patient due to the less number of unsuccessful punctures.

For the calculation of the required sample, since the incidence of our primary end-point of a compound of crossover to femoral access and/or access site-related vascular complications has not been reported so far, the sample will be calculated with the rate of events obtained in our center at 6 months of recruiting patients. For this calculation, the proportional difference formula with an alpha value of 0,05 and a beta value of 0,20 will be used to have a statistical power of 80%. The investigators estimate that 1,500 patients will be required in a 11-month period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years, scheduled consecutively to perform a coronary procedure in the department of hemodynamics of the National Institute of Cardiology "Ignacio Chavez".
* Patients may have any of the following indications for cardiac catheterization: Thoracic pain under study. Stable chronic coronary disease. Acute myocardial infarction with ST segment elevation, not perfused (without timely reperfusion therapy) with less than 4 weeks of evolution. Acute myocardial infarction with ST-segment elevation, successful thrombolytic therapy, which will undergo drug-invasive therapy. Acute myocardial infarction without ST segment elevation. Unstable angina. Any acute coronary syndrome, to intervene non-infarct-related artery. Disease of any heart valve. Myocarditis or pericarditis. Dilated cardiomyopathy. Patients in renal or cardiac transplantation protocol for any etiology. Congenital heart disease that requires knowing the coronary anatomy prior to surgical correction.
* The planned procedure can be any of the following: For diagnostic purposes (coronary angiography only, left catheterization, left and right catheterization). For therapeutic purposes: percutaneous coronary intervention (PCI), with or without stent placement.
* A priori access must be right or left radial artery.
* Radial arterial pulse may be present or absent by palpation.
* Modified Allen or Barbeau test should be positive (presence of collateral palmar flow).

Exclusion Criteria:

* Pregnant.
* Not have informed consent for the present clinical trial, or do not fully understand the meaning of informed consent.
* With acute myocardial infarction with ST segment elevation in the first 12 hours from the onset of symptoms.
* With any acute coronary syndrome complicated with acute pulmonary edema, cardiogenic shock and / or malignant ventricular arrhythmias.
* In which a cardiac catheterization is planned a priori to be performed via femoral, brachial or ulnar.
* Patients in whom first attempt of arterial puncture is performed by 2nd year interventional cardiology fellow or by physician in charge.
* Participating in another clinical trial.
* Be allergic or have contraindications to nitroglycerin or other nitrates.
* Any phosphodiesterase 5 inhibitor (sildenafil, tadalafil, avanafil, vardenafil) has been taken within 72 hours prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
Compound of crossover to femoral access and/or access site-related vascular complications. | Within 72 hours or at hospital discharge (whichever occurs first).
  Crossover to femoral access: number of cases in which the procedure could not be completed via radial artery and access via femoral artery was changed. Access site-related vascular complications: hematoma requiring intervention as an additional compression bandage, radial perforation / dissection, hemorrhage requiring transfusion, compartment syndrome, arteriovenous fistula, pseudoaneurysm, or any complication requiring surgical intervention.

SECONDARY OUTCOMES:
Number of attempts to cannulate the radial artery (punctures). | Through study completion, an average of 1 year.
  Number of times the needle is inserted through the skin with the intention of puncturing the radial artery. This outcome measure will be assessed by interventional cardiology fellow who applies the maneuver and attempt to cannulate the artery.
Time until obtaining the radial access. | Through study completion, an average of 1 year.
  Counted from the first attempt to puncture the radial artery, from the needle through the skin to the successful insertion of the introducer into the radial artery with adequate blood return.
Improvement in radial pulse strength. | Through study completion, an average of 1 year.
  The interventional cardiologist fellow who will apply the maneuver, will assess the strength of the radial pulse before the administration of the maneuver and at least 1 minute after, and will record the change in pulse strength. Pulse Score: 0 - No palpable pulse. 1 - Weak pulse. 2 - Pulse of normal intensity. 3 - Very intense pulse.
Loss of radial artery flow (radial artery occlusion) at 30 days. | At 30 days.
  The maximum longitudinal and transverse diameter of the radial artery and the maximum arterial flow velocity will be measured, with the transducer placed 1 cm proximal to the styloid process using ultrasound doppler with a vascular transducer.
Pain in the cannulated extremity. | Through study completion, an average of 1 year.
  It will be evaluated with a visual-analogue subjective pain scale from 1 to 10 referred by the patient. Pain will be assessed at the time of introducing the radial introducer.
Radial spasm. | During coronary procedure.
  It will be referred to as radial spasm if the patient reports pain or discomfort of any intensity at the cannulated end, at the time of manipulating, advancing and / or withdrawing any catheter through the arterial introducer. Angiographic confirmation of spasm may or may not be done. Additional intra-arterial vasodilators, or additional IV analgesics, may or may not be administered at the discretion of the operator.
Headache. | During coronary procedure.
  Referred by the patient during any time of the procedure in the hemodynamic laboratory. It will be recorded on a subjective-to-analogue subjective pain scale from 1 to 10.
Hypotension. | In the following 10 minutes after administration of the maneuver.
  Systolic blood pressure lower than 90 mmHg in the following 10 minutes after the maneuver, not related to the manipulation of a coronary artery with any device.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Peña Duque, MD, Study Director — Director of Department of Interventional Cardiology, National Institute of Cardiology, Mexico City, Mexico.
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
I will show the IPD during my research seminar wich is part of the program to being doctor in medical sciences to obtain a PhD degree.